CLINICAL TRIAL: NCT02472522
Title: Comparative Study of Ropivacaine and Ropivacaine With Dexmeditomedine in Transversus Abdominis Plane (TAP) Block for Post-operative Analgesia in Patients Undergoing Cesarean Sections
Brief Title: Comparative Study of Ropivacaine and Ropivacaine With Dexmeditomedine in TAP Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Main Hospital (Other)
Responsible Party: Principal Investigator, Dr.Deb Sanjay Nag, Associate Specialist, Tata Main Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SR9851450
Record Dates: First submitted 2015-06-09; First posted 2015-06-16 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-05

CONDITIONS: Pregnancy
MeSH Terms: interventions — Ropivacaine; Dexmedetomidine; Adrenergic Agonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Placebo Comparator): Patients satisfying inclusion criteria will receive Subarachnoid Block with Bupivacaine Heavy 0.5% (11 mg/2.2 ml) with 25 micrograms of fentanyl. At the end of the procedure, bilateral TAP block will be performed using Landmark Technique with 2.5 mg/kg of ropivacaine diluted with 0.9% saline to a total volume of 40 ml (20 ml each side)
  Interventions: Other: Ropivacaine
- Ropivacaine + Dexmedetomidine (Experimental): Patients satisfying inclusion criteria will receive Subarachnoid Block with Bupivacaine Heavy 0.5% (11 mg/2.2 ml) with 25 micrograms of fentanyl. At the end of the procedure, bilateral TAP block will be performed using Landmark Technique with addition of Dexmedetomidine 1 micrograms/kg to with 2.5 mg/kg of ropivacaine diluted with 0.9% saline to a total volume of 40 ml (20 ml each side) for the TAP block
  Interventions: Drug: Ropivacaine + Dexmedetomidine

INTERVENTIONS:
Drug: Ropivacaine + Dexmedetomidine — Patients satisfying inclusion criteria will receive Subarachnoid Block with Bupivacaine Heavy 0.5% (11 mg/2.2 ml) with 25 micrograms of fentanyl. At the end of the procedure, bilateral TAP block will be performed using Landmark Technique with 2.5 mg/kg of ropivacaine and 1 micrograms/kg dexmedetomidine (combination drug) diluted with 0.9% saline to a total volume of 40 ml (20 ml each side) for the TAP block
  Other Names: selective alpha 2 (α2) adrenergic agonist
  Arms: Ropivacaine + Dexmedetomidine
Other: Ropivacaine — Patients satisfying inclusion criteria will receive Subarachnoid Block with Bupivacaine Heavy 0.5% (11 mg/2.2 ml) with 25 micrograms of fentanyl. At the end of the procedure, bilateral TAP block will be performed using Landmark Technique with 2.5 mg/kg of ropivacaine diluted with 0.9% saline to a total volume of 40 ml (20 ml each side)
  Arms: Ropivacaine

SUMMARY:
Comparative study of Ropivacaine and Ropivacaine with dexmedetomidine in transversus abdominis plane (TAP) block for post-operative analgesia in patients undergoing Caesarean Section.

DETAILED DESCRIPTION:
Patients satisfying inclusion criteria will receive Subarachnoid Block with Bupivacaine Heavy 0.5% (11 mg/2.2 ml) with 25 micrograms of fentanyl. Routine NPO protocols will be followed. At the end of the procedure, bilateral TAP block will be performed using Landmark Technique in Triangle of Petit with 2 inches 24 G needle.

Patients would receive 75 mg of intramuscular diclofenac sodium immediately on shifting to the postoperative care unit (PACU) and a second dose 12 hours later. The time after the TAP block when rescue analgesia was first sought, total dose of required morphine in 24 hours postoperatively, its adverse effects like pruritus, nausea and vomiting will be recorded. VAS will be used to assess post-operative pain (VAS; where 0 = no pain and 10 = worst imaginable pain) during rest and on coughing.

Rescue analgesia would be provided with 6 mg of intravenous morphine and additional doses of 3 mg at 10 minutes interval till VAS was less than 3 or in case of development of adverse effects such as nausea and/or vomiting, respiratory depression (SpO2 <92%, ventilatory frequency rate <10), or occurrence of deep sedation (eyes closed >3 min, Ramsay Score RS >2). An RS on a 6-point scale was used (1=anxious and agitated patient; 2=cooperative patient; 3=asleep patient, brisk response to loud voice; 4=asleep patient, sluggish response to loud voice; 5=no response to loud voice; score of 6=no response to pain). In PACU and in first 24 h post-operatively, MAP, HR, VAS (at rest and on coughing), nausea and vomiting, sedation score (RS) will be recorded on admission to PACU and at 1,4, 8, 12, 18 and 24 hours post-operatively by an observer who will be unaware of the study protocol.

Patients will we assessed on a 5 point scale at the end of 24 hours on the quality of postoperative analgesia. Nausea and vomiting will be recorded using a categorical scoring system (0 = none, 1 = nausea, 2 = retching, 3 = vomiting). IV Metoclopramide 10 mg bolus will be offered for any patient with a score >/=1.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2
* Age above 18 years
* Patients for Lower Section Cesarean Section surgery

Exclusion Criteria:

* Patient refusal
* Allergy to study medications
* Localized infection over injection point
* Patients with significant coagulopathies and with contraindications to regional anesthesia
* Patients with a history of cardiac, respiratory, renal or hepatic failure
* Psychological disorders
* Chronic use of pain medications or adrenoreceptors agonists or antagonists.
* BMI >35 or weight < 50 kilograms

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priti Gehlot, DA, Principal Investigator — Tata Main Hospital, Jamshedpur, India
Locations (1):
- Tata Main Hospital, Jamshedpur, Jharkhand, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between May 2015 to November 2015 in the Obstetrics and Gynaecology Operation Theater and Post-operative ward of the Tata Main Hospital, Jamshedpur, India.
Groups:
- Ropivacaine + Dexmedetomidine: Patients satisfying inclusion criteria will receive Subarachnoid Block with Bupivacaine Heavy 0.5% (11 mg/2.2 ml) with 25 micrograms of fentanyl. At the end of the procedure, bilateral TAP block will be performed using Landmark Technique with addition of Dexmedetomidine 1 micrograms/kg to with 2.5 mg/kg of ropivacaine diluted with 0.9% saline to a total volume of 40 ml (20 ml each side) for the TAP block
  Ropivacaine + Dexmedetomidine: Addition of Dexmedetomidine 1 micrograms/kg (to with 2.5 mg/kg of ropivacaine diluted with 0.9% saline to a total volume of 40 ml ) for the TAP block
Period: Overall Study
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with term pregnancy who were posted for Lower segment caesarean section were recruited for the study
Groups:
- Ropivacaine: Patients satisfying inclusion criteria will receive Subarachnoid Block with Bupivacaine Heavy 0.5% (11 mg/2.2 ml) with 25 micrograms of fentanyl. At the end of the procedure, bilateral TAP block was performed using Landmark Technique with 2.5 mg/kg of ropivacaine diluted with 0.9% saline to a total volume of 40 ml (20 ml each side)
  Ropivacaine: Patients satisfying inclusion criteria will received Subarachnoid Block with Bupivacaine Heavy 0.5% (11 mg/2.2 ml) with 25 micrograms of fentanyl. At the end of the procedure, bilateral TAP block will be performed using Landmark Technique with 2.5 mg/kg of ropivacaine diluted with 0.9% saline to a total volume of 40 ml (20 ml each side)
- Ropivacaine + Dexmedetomidine: Patients satisfying the inclusion criteria received Subarachnoid Block with Bupivacaine Heavy 0.5% (11 mg/2.2 ml) with 25 micrograms of fentanyl. At the end of the procedure, bilateral TAP block was performed using Landmark Technique with addition of Dexmedetomidine 1 micrograms/kg to with 2.5 mg/kg of ropivacaine diluted with 0.9% saline to a total volume of 40 ml (20 ml each side) for the TAP block
  Ropivacaine + Dexmedetomidine: Addition of Dexmedetomidine 1 micrograms/kg (to with 2.5 mg/kg of ropivacaine diluted with 0.9% saline to a total volume of 40 ml ) for the TAP block
- Total: Total of all reporting groups
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.02 (4.64) | 28.66 (4.53) | 28.34 (4.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 50 | 50 | 100
Weight [Mean (Standard Deviation); unit: Kilograms] | 64.08 (5.96) | 65.68 (7.49) | 64.88 (6.78)
Height of the patients [Mean (Standard Deviation); unit: Centimeters] | 158.90 (4.53) | 157.36 (15.77) | 158.13 (11.57)
Duration of surgery [Mean (Standard Deviation); unit: Minutes] | 50.12 (3.97) | 50.00 (4.35) | 50.06 (4.14)

OUTCOME MEASURES:

1. Primary Outcome: The Time After the TAP Block When Rescue Analgesia Was First Sought
Time Frame: 24 hours
Population: Number of patients who sought rescue analgesic within the first 24 hours postoperatively. Rest of the studied patients needed no rescue analgesic within the first 24 hours postoperatively.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 25 | 14
Hours | 13.12 (3.53) | 18.21 (3.14)

2. Secondary Outcome: Total Dose of Required Morphine in 24 Hours Postoperatively
Time Frame: 24 hours
Population: Only the mentioned number of patients needed analgesia within the first 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 25 | 14
Milligrams | 8.16 (2.94) | 6.21 (0.8)

3. Secondary Outcome: Adverse Effects Like Pruritus, Nausea and Vomiting
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
participants
  Nausea | 1 | 0
  Vomiting | 2 | 1
  No adverse effect | 47 | 49

4. Other Pre Specified Outcome: Mean Arterial Pressure (MAP): Intraoperative Period
Description: The Mean Arterial Pressure (MAP) of the patients were recorded from the start of surgery up to 60 minutes at 5, 10, 20, 30, 40, 50, 60 mins. No surgery lasted more than 60 minutes.
Time Frame: Upto 60 minutes
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
millimeter of mercury (mmHg)
  Baseline | 76.84 (8.57) | 79.38 (10.40)
  At 5 minutes | 68.28 (7.90) | 66.38 (7.97)
  At 10 minutes | 67.42 (6.26) | 67.52 (8.62)
  At 20 minutes | 70.02 (7.24) | 68.98 (8.63)
  At 30 minutes | 72.46 (7.39) | 73.44 (8.68)
  At 40 minutes | 75.82 (7.93) | 77.76 (9.55)
  At 50 minutes | 76.98 (8.89) | 79.90 (10.67)
  At 60 minutes | 79.66 (10.10) | 84.02 (12.94)

5. Other Pre Specified Outcome: Heart Rate: Intraoperative Period
Description: The Heart Rate of the patients were recorded from the start of surgery up to 60 minutes at 5, 10, 20, 30, 40, 50, 60 mins. No surgery lasted more than 60 minutes.
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
beats/minute
  Baseline | 85.64 (7.75) | 86.76 (9.54)
  At 5 minutes | 94.52 (10.68) | 98.20 (11.54)
  At 10 minutes | 96.60 (11.92) | 97.02 (11.75)
  At 20 minutes | 93.84 (10.35) | 93.28 (10.46)
  At 30 minutes | 91.08 (8.71) | 90.06 (9.99)
  At 40 minutes | 87.96 (8.46) | 88.68 (10.24)
  At 50 minutes | 86.60 (8.84) | 87.52 (10.17)
  At 60 minutes | 86.74 (9.44) | 88.50 (11.28)

6. Other Pre Specified Outcome: Time to Complete Disappearance of Motor Block
Description: During the postoperative recovery, the level of motor block was assessed with Modified Bromage Scale 0 = no paralysis, able to flex hips/knees/ankles
  1. = able to move knees, unable to raise extended legs
  2. = able to flex ankles, unable to flex knees
  3. = unable to move any part of the lower limb The time from subarachnoid block to complete disappearance of motor block (Bromage 0) was recorded in minutes.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
minutes | 171.06 (5.51) | 170.34 (14.62)

7. Other Pre Specified Outcome: Duration of Sensory Loss at T10 Level
Description: The duration of sensory loss (from the subarachnoid block) at T10 level was assessed by pin-prick test by a sterile needle in minutes.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
minutes | 303.74 (7.86) | 305.40 (7.19)

8. Other Pre Specified Outcome: Mean Arterial Pressure (MAP): Postoperative Period
Description: The Mean Arterial Pressure (MAP) of the patients were recorded after shifting from Operation Theater and at 1, 4, 8,12,18 and 24th hour after shifting to the postoperarive area.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
millimeter of mercury (mmHg)
  On shifting | 79.98 (10.13) | 83.80 (13.33)
  1 hour | 80.14 (10.58) | 83.46 (12.13)
  4 hours | 78.38 (9.72) | 82 (11.60)
  8 hours | 78.06 (8.34) | 81.26 (10.65)
  12 hours | 82.90 (10.64) | 80.84 (9.80)
  18 hours | 83.94 (7.07) | 85.08 (13.89)
  24 hours | 77.24 (5.64) | 79.46 (7.76)

9. Other Pre Specified Outcome: Heart Rate: Postoperative
Description: The Heart Rate of the patients were recorded after shifting from Operation Theater and at 1, 4, 8,12,18 and 24th hour after shifting to the postoperarive area.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
beats/minute
  On shifting | 84.92 (13.90) | 88.52 (12.59)
  At 1 hour | 86.74 (9.56) | 86.50 (12.09)
  At 4 hours | 83.50 (8.07) | 82.54 (10.01)
  At 8 hours | 81.46 (9.11) | 81.14 (10.00)
  At 12 hours | 85.26 (13.48) | 83.18 (8.03)
  At 18 hours | 80.88 (10.44) | 81.60 (15.52)
  At 24 hours | 78.82 (6.59) | 79.14 (6.64)

10. Other Pre Specified Outcome: Visual Analogue Scale at Rest (VAS-R)
Description: Visual Analogue Scale at rest (VAS-R) was used to assess Post-operative Pain at rest. Where: 0 = no Pain and 10 = Worst Imaginable Pain. They were Recorded on Shifting to Postoperative and Then at 1, 4, 8, 12, 18 and 24 Hour
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
Units on a scale
  On shifting to postoperative area | 0.06 (0.31) | 0.00 (0.0)
  At 1 hour | 0.36 (0.56) | 0.38 (0.53)
  At 4 hours | 0.94 (0.65) | 0.96 (0.53)
  At 8 hours | 1.46 (0.86) | 1.34 (0.74)
  At 12 hours | 2.54 (1.49) | 1.66 (0.52)
  At 18 hours | 2.74 (1.44) | 2.12 (0.72)
  At 24 hours | 1.88 (0.38) | 1.78 (0.42)

11. Other Pre Specified Outcome: Visual Analogue Scale on Coughing (VAS-C)
Description: Visual Analogue Scale on Coughing (VAS-C) Was Used to Assess Post-operative Pain on Coughing. Where: 0 = no Pain and 10 = Worst Imaginable Pain. They were Recorded on Shifting to Postoperative and Then at 1, 4, 8, 12, 18 and 24 Hour
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
Units on a scale
  On shifting to postoperative area | 0.24 (0.52) | 0.08 (0.27)
  At 1 hour | 1.12 (0.75) | 0.96 (0.57)
  At 4 hours | 1.58 (0.70) | 1.48 (0.54)
  At 8 hours | 2.22 (1.05) | 1.94 (0.65)
  At 12 hours | 3.42 (1.76) | 2.40 (0.64)
  At 18 hours | 3.52 (1.49) | 3.02 (0.82)
  At 24 hours | 2.62 (0.60) | 2.64 (0.52)

12. Other Pre Specified Outcome: Short Assessment of Patient Satisfaction Score (SAPS)
Description: Short assessment of patient satisfaction score(SAPS) was assessed on a 5 point scale at the end of 24 hours on the quality of postoperative analgesia. where:
  1. highly dissatisfied
  2. dissatisfied
  3. neither dissatisfied nor satisfied
  4. satisfied
  5. highly satisfied
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
Units on a scale | 4.22 (0.93) | 4.70 (0.50)

13. Post Hoc Outcome: Percentage of Patients Needing Rescue Analgesic
Description: Percentage of patients needing rescue analgesic. Rescue analgesia was provided with 6 mg of intravenous morphine and additional doses of 3 mg at 10 minutes interval till VAS was less than 3 or the development of adverse effects such as nausea and/or vomiting, respiratory depression (SpO2 <92%, ventilatory frequency rate <10), or occurrence of deep sedation (eyes closed >3 min, Ramsay Score RS >2).
Time Frame: 24 hours
Measure: Number; unit: percentage needing rescue analgesic
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Number analyzed (Participants) | 50 | 50
percentage needing rescue analgesic | 50 | 28

ADVERSE EVENTS:
Time Frame: 1st 24 hours postoperatively
Arm/Group | Ropivacaine | Ropivacaine + Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 3/50 | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropivacaine (N=50) | Ropivacaine + Dexmedetomidine (N=50)
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
1. There was no mechanism in our study to ascertain the effectiveness or failure of the TAP block.
2. We did not ascertain if the effect of dexmedetomidine was by its systemic absorption or by a perineural effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No